CLINICAL TRIAL: NCT04323007
Title: Thyroid Dysfunction in Patients With Nephrotic Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Merna Makram (Other)
Collaborators: Assiut University (Other)
Responsible Party: Sponsor-Investigator, Merna Makram, Thyroid Dysfunction in patients with nephrotic syndrome, Assiut University
Organization: Assiut University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Thyroid Dysfunction
Record Dates: First submitted 2020-01-12; First posted 2020-03-26 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Thyroid Dysfunction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nephrotic syndrome patients (Other): This study is to evaluate Thyroid Hormone profile in patients with Nephrotic syndrome to identify clinical predictor of Thyroid dysfunction in patients with Nephrotic syndrome
  Interventions: Diagnostic Test: Nephrotic patients

INTERVENTIONS:
Diagnostic Test: Nephrotic patients — Laboratory measures will include Blood sugar Urine analysis with 24hrs protein in urine Complete blood count Liver function tests Kidney functions test Plasma lipid levels Thyroid functions test Abdominal ultrasound Antithyrperoxidase Renal biopsy

SUMMARY:
This study is to evaluate Thyroid Hormone profile in patients with Nephrotic syndrome to identify clinical predictor of Thyroid dysfunction in patients with Nephrotic syndrome

DETAILED DESCRIPTION:
Nephrotic syndrome (NS) is one of the most popular glomerular diseases all over the world It result in loss of various macromolecules which exist in the plasma and bound to plasma proteins. They are carried away and lost in the urine due to increase glomerular membrane permeability.The abnormalities arising as a result of persistence of generalized edema , substantial heavy proteinuria >3,5 gm/24 h 3, hypoalbuminemia<30 g/L and hyperlipidemia Also, nephrotic syndrome may associated with thromboembolism and increase risk of infection, vitamin D deficiency, Iron deficiency and endocrine abnormalities such as primary Hypothyroidism.The interaction between kidney and Thyroid hormone is an important factor in the normal functioning of both the vital organs, thyroid hormone play a major role in early development of kidney structurally and regulation of major glomerular and tubular function and water and electrolytes balance .Kidneys on other hand are important in the metabolism and elimination of Thyroid Hormone.The effect of nephrotic syndrome on thyroid function can be explained by presence of proteinuria and loss of Thyroid binding globulins (TBG) in urine

which lead to decrease in Total T3,Total T4,free T3 and free T4 and consequently increase in TSH from the pituitary gland with over function of thyroid gland in order to maintain Thyroid hormone levels. Another theory explain association between nephrotic syndrome and thyroid dysfunction is Autoimmunity which can attack both organs and may also cause abnormal function of both organs. Thus, subclinical Hypothyroidism and overt Hypothyroidism may happen in NS patients and CKD patients

ELIGIBILITY:
Inclusion Criteria:

* Nephrotic syndrome defined by the following:

  1. Generalized edema
  2. Urine protein excretion > 3,5 g/24 hours
  3. Urine protein to creatinine ratio > 3,500mg/g
  4. Serum albumin level less than 30 g/L

Exclusion Criteria:

- 1) Patients < 18 years old 2) Patients who have Thyroid diseases, current or past history of thyroid hormone or antithyroid drug intake.

3) Patients who have diabetes mellitus or autoimmune diseases as systemic lupus erythematosus and RA 4) Medications known to affect thyroid function. 5) Patients with liver cirrhosis and chronic liver disease as augmentin

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Hypothyroidism in patients with nephrotic syndrome | 1year
  Decrease T3 and/or T4 and/or increase TSH in patients with proteinurea more than 3.5 mg

REFERENCES:
- [Background] McCloskey O, Maxwell AP. Diagnosis and management of nephrotic syndrome. Practitioner. 2017 Feb;261(1801):11-5. PMID 29020719
- [Background] Bradley SE, Stephan F, Coelho JB, Reville P. The thyroid and the kidney. Kidney Int. 1974 Nov;6(5):346-65. doi: 10.1038/ki.1974.119. No abstract available. PMID 4431166